CLINICAL TRIAL: NCT05387161
Title: Evaluation of Nutritional Status, Eating Habits and Improvement of Symptoms With a Nutritional Intervention in Women With enDometriosis and chrOnic Pelvic Pain
Brief Title: Evaluation of Nutritional Status, Eating Habits and Improvement of Symptoms With a Nutritional Intervention in Women With enDometriosis
Acronym: ENDO-DIET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Pavia (Other)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Cinzia Ferraris, Researcher, University of Pavia
Other Study IDs: 2021-ENDODIET
Record Dates: First submitted 2022-01-24; First posted 2022-05-24 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Endometriosis
Keywords: endometriosis; diet; inflammation; chronic pelvic pain
MeSH Terms: conditions — Endometriosis; Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: A nutritional assessment will be held with the detection of anthropometric parameters. Each participant will be asked to fill in the SF36, the VAS scales, the KESS questionnaire, the SFFI questionnaire, the Questionnaire PUF and O'Leary/Santn, the BDI and the TAS for an assessment of the psychological component.
  In addition, patients will be asked to fill in a FFQ of food consumption and a 7 days food diary. Finally, routine blood chemistry tests will also be performed, to which will be added those for measuring the inflammatory state and stool examination for the evaluation of fecal Calprotectin for the measurement of intestinal inflammatory markers.
  The nutritional intervention will consist in providing general nutritional indications specific for endometriosis and an indicative daily diet plan, which must be followed for 6 months.
  At the end of the 6 months, all anthropometric assessments, blood chemistry and stool tests will be repeated, together with the questionnaires.
  Interventions: Other: Nutritional intervention

INTERVENTIONS:
Other: Nutritional intervention — The nutritional intervention will consist in providing general nutritional indications specific for endometriosis and an indicative ungrammatical daily diet plan, which must be followed for the entire period of intervention (6 months).

SUMMARY:
The study aims to investigate the nutritional status and eating habits of women suffering from endometriosis and chronic pelvic pain in relation to describe the possible improvement of clinical symptoms following a nutritional intervention.

The primary aim is to describe and evaluate the impact of nutritional intervention on clinical symptoms (pain, quality of life and intestinal function) in women suffering from endometriosis with chronic pelvic pain.

The first secondary aim will be to describe and evaluate the impact of the nutritional intervention by describing the changes in some specific areas of the patients (sexual, psychological) together with the quantification of some routine blood chemistry parameters (inflammatory markers, levels of proteins and vitamins) .

The second secondary objective will be aimed at describing the changes in clinical symptoms and the parameters mentioned above in patients based on the severity/stage of the pathologies under study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of endometriosis +/- chronic pelvic pain
* No menopause (at least 1 menstrual cycle in the previous 6 months)
* Informed consent from the patient and / or an authorized legal representative

Exclusion Criteria:

* Postmenopause
* Pregnancy
* Hysterectomy or oophorectomy
* Chronic diseases that affect the gastrointestinal absorption of nutrients (celiac disease, Chron's disease, ulcerative colitis, cystic fibrosis)
* History of kidney stones, cancer (except basal cell carcinoma) or diabetes
* Modification in the course of the therapeutic intervention of the therapy for endometriosis

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients referred to the Endometriosis Outpatient Clinic of the Gynecological Clinic of the San Matteo Polyclinic in Pavia will be enrolled and will agree to participate in the study and have signed the relative informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is to describe and evaluate the impact of nutritional intervention on clinical symptoms (pain, quality of life and intestinal function) in women suffering from endometriosis with chronic pelvic pain. | 6 months
  The outcome will be assessed with repeated measurements using the following parameters:
  -Evaluation of chronic pelvic pain, dysmenorrhea, dyschezia and dysuria: VAS visual analogue scale, from 0 to 10 points where 10 points indicates worst pain
The primary outcome is to describe and evaluate the impact of nutritional intervention on clinical symptoms (quality of life) in women suffering from endometriosis with chronic pelvic pain. | 6 months
  The outcome will be assessed with repeated measurements using the following parameters:
  Quality of life: measurement of physical and mental components with SF36 consisting of two components, one physical and one mental. Both fall within a range from 0 to 100 points where higher values are associated with better health
The primary outcome is to describe and evaluate the impact of nutritional intervention on clinical symptoms (intestinal function) in women suffering from endometriosis with chronic pelvic pain. | 6 months
  The outcome will be assessed with repeated measurements using the following parameters:
  Bowel Function: Knowles-Eccersley-Scott Symptom Questionnaire (KESS) (points)

SECONDARY OUTCOMES:
The secondary outcome will be to describe and evaluate the impact of the nutritional intervention by describing the changes in Sexual Function | 6 months
  The outcomes necessary to respond to the secondary objective are the administration of the following questionnaire:
  Sexual Function: FSFI questionnaire (points)
To describe and evaluate the impact of the nutritional intervention by describing the changes in Urinary function and bladder pain | 6 months
  The outcomes necessary to respond to the secondary objective are the administration of the following questionnaire:
  Urinary function and bladder pain: PUF and O's Leary / Sant questionnaire (points)
The secondary outcome will be to describe and evaluate the impact of the nutritional intervention by describing the changes in Psychological component about Depression | 6 months
  The outcomes necessary to respond to the secondary objective are the administration of the following questionnaire:
  Beck Depression Inventory (BDI) (points)
The secondary outcome will be to describe and evaluate the impact of the nutritional intervention by describing the changes in Psychological component | 6 months
  The outcomes necessary to respond to the secondary objective are the administration of the following questionnaires:
  Alexithymia Scale (TAS) questionnaire (points)
The secondary outcome will be to describe and evaluate the impact of the nutritional intervention by describing the changes in some routine blood chemistry parameters | 6 months
  The outcomes necessary to respond to the secondary objective are the administration of the following routine blood chemistry parameters:
  Measure Ca125 (unità/ml) and Vitamin D (ng/ml)
The secondary outcome will be to describe and evaluate the impact of the nutritional intervention by describing the changes in Intestinal inflammatory marker | 6 months
  The outcomes necessary to respond to the secondary objective are the administration of the following test:
  fecal calprotectin (mg/kg)
The secondary outcome will be to describe and evaluate the impact of the nutritional intervention by describing the changes in some Inflammatory markers | 6 months
  The outcomes necessary to respond to the secondary objective are the administration of the following Inflammatory markers: IL-6 and IL-1β values (pg/ml)
The secondary outcome will be to describe and evaluate the impact of the nutritional intervention by describing the changes in measurement of proteins | 6 months
  The outcomes necessary to respond to the secondary objective are the administration of the following measurement of proteins: C-reactive protein values (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Gardella, Dott, Study Director — IRCCS Policlinico San Matteo
Locations (1):
- University of Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No